CLINICAL TRIAL: NCT07083440
Title: A Clinical Investigation of Varied Remimazolam Dosages With Sufentanil and Propofol for Painless Pediatric Gastrointestinal Endoscopy
Brief Title: Varied Remimazolam Dosages for Pediatric Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Hebei Province (Other)
Responsible Party: Principal Investigator, Wenjing Chen, Principal investigator, Children's Hospital of Hebei Province
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECH-2023-010
Record Dates: First submitted 2025-06-19; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Diseases
Keywords: Remimazolam; Painless gastrointestinal endoscopy; Sufentanil; Propofol; Pediatric
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — remimazolam; Propofol; Sufentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam 0.2 mg/kg Group (R2) (Experimental): Experimental. Patients receive remimazolam 0.2 mg/kg.
  Interventions: Drug: Remimazolam; Drug: Propofol; Drug: Sufentanil
- Remimazolam 0.3 mg/kg Group (R3) (Experimental): Experimental. Patients receive remimazolam 0.3 mg/kg.
  Interventions: Drug: Remimazolam; Drug: Propofol; Drug: Sufentanil
- Remimazolam 0.4 mg/kg Group (R4) (Experimental): Experimental. Patients receive remimazolam 0.4 mg/kg.
  Interventions: Drug: Remimazolam; Drug: Propofol; Drug: Sufentanil

INTERVENTIONS:
Drug: Remimazolam — Intravenous bolus administered over 1 minute (prepared as a 1 mg/mL solution). Doses: 0.2 mg/kg, 0.3 mg/kg, or 0.4 mg/kg according to group allocation.
Drug: Propofol — Intravenous (10 mg/mL emulsion), initial titrated dose ranging from 0.5 to 2 mg/kg, administered slowly until MOAA/S ≤ 2. Supplemental 0.5 mg/kg boluses as needed.
Drug: Sufentanil — Intravenous dose of 0.1 µg/kg administered approximately 30 minutes before the start of the procedure.

SUMMARY:
This prospective, randomized, comparative study aims to compare the efficacy and safety of three different doses of remimazolam (0.2 mg/kg, 0.3 mg/kg, and 0.4 mg/kg) combined with sufentanil and propofol for painless gastroscopy in pediatric patients. The study will assess sedation quality, propofol consumption, hemodynamic stability, and adverse event profiles to identify an optimal remimazolam dosing regimen.

DETAILED DESCRIPTION:
Pediatric patients undergoing gastrointestinal endoscopy often require deep sedation. Propofol is commonly used but can cause injection pain, respiratory depression, and hemodynamic instability. Remimazolam, a novel ultra-short-acting benzodiazepine, offers rapid onset, predictable recovery, and potentially better hemodynamic stability. This study investigates three doses of remimazolam (0.2 mg/kg, 0.3 mg/kg, and 0.4 mg/kg) co-administered with sufentanil (0.1 µg/kg) and titrated propofol to achieve a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤ 2 in 180 pediatric patients (ASA I-II, aged <18 years) undergoing gastroscopy. Patients are randomly assigned to one of three remimazolam dose groups. The study will evaluate total propofol dosage, hemodynamic changes (blood pressure, heart rate), time to sedation, awakening and recovery times, incidence of adverse events (e.g., hypotension, respiratory depression, injection pain), and satisfaction scores. The goal is to determine a remimazolam dose that provides effective sedation with reduced propofol requirements and an improved safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective gastrointestinal endoscopy under anesthesia.
* Patients classified as American Society of Anesthesiologists (ASA) physical status I or II.
* Patients aged 3 to under 18 years of age.
* Written informed consent provided by parents or legal guardians.

Exclusion Criteria:

* Patients with known or suspected difficult airway, severe systemic disease (ASA ≥ III).
* Uncorrected significant abnormal liver or kidney function that could significantly alter drug metabolism (e.g., AST/ALT > 2x upper limit of normal, eGFR < 30 mL/min/1.73m²).
* Known allergy to study medications (remimazolam, propofol, sufentanil, or their components including egg or soy for propofol).
* Congenital illnesses such as severe congenital heart disease, or other conditions that may impact treatment observation or increase anesthetic risk.
* Patients who were obese (defined as BMI > 95th percentile for age and sex) or severely malnourished (BMI < 3rd percentile for age and sex).
* Patients who had taken sedatives, opioid analgesics (other than prescribed for chronic pain), or psychotropic medications (e.g., antidepressants, antipsychotics) within 24 hours prior to the procedure (unless part of their regular, stable medication regimen for a chronic condition, as assessed and deemed safe by the anesthesiologist).
* Patients with pre-existing severe, uncontrolled mental illness or significant cognitive dysfunction that would preclude assessment of sedation or cooperation.
* Patients who had participated in other clinical trials within the past 4 weeks.
* Contraindications to the planned endoscopic procedure (e.g., recent gastrointestinal perforation, bowel obstruction).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Total Propofol Dosage | Periprocedural (during the gastroscopy procedure, lasting approximately 15-30 minutes)
  Total amount of propofol (mg) administered during the gastroscopy procedure to maintain MOAA/S score ≤ 2.
Incidence of Hypotension | From induction of anesthesia through discharge from the Post-Anesthesia Care Unit (up to approximately 2 hours)
  Percentage of patients experiencing hypotension, defined as a systolic blood pressure (SBP) decrease greater than 20% from baseline or below the 5th percentile for age, sustained for >2 minutes, or requiring intervention.

SECONDARY OUTCOMES:
Hemodynamic Stability: Systolic Blood Pressure (SBP) | From Baseline through discharge from the Post-Anesthesia Care Unit (up to approximately 2 hours post-procedure).
  Systolic Blood Pressure (SBP) in mmHg. Assessed at 6 time points: Baseline (before anesthesia induction), immediately after induction, at gastroscope insertion, 5 minutes after gastroscope insertion, upon patient awakening, and at discharge from the Post-Anesthesia Care Unit (PACU).
Hemodynamic Stability: Diastolic Blood Pressure (DBP) | From Baseline through discharge from the Post-Anesthesia Care Unit (up to approximately 2 hours post-procedure).
  Diastolic Blood Pressure (DBP) in mmHg. Assessed at 6 time points: Baseline (before anesthesia induction), immediately after induction, at gastroscope insertion, 5 minutes after gastroscope insertion, upon patient awakening, and at discharge from the Post-Anesthesia Care Unit (PACU).
Hemodynamic Stability: Heart Rate (HR) | From Baseline through discharge from the Post-Anesthesia Care Unit (up to approximately 2 hours post-procedure).
  Heart Rate (HR) in beats/minute. Assessed at 6 time points: Baseline (before anesthesia induction), immediately after induction, at gastroscope insertion, 5 minutes after gastroscope insertion, upon patient awakening, and at discharge from the Post-Anesthesia Care Unit (PACU).
Success Rate of Sedation | At the conclusion of the gastroscopy procedure
  Percentage of patients successfully completing gastroscopy with MOAA/S ≤ 2 without requiring alternative sedative agents or premature termination.
Time to Induce Sedation | During the induction of anesthesia (within the first 5 minutes)
  Time (minutes) from start of remimazolam injection to MOAA/S ≤ 2.
Awakening Time | Immediately following the end of the procedure
  Time (minutes) from the last dose of sedative/end of procedure to the patient opening their eyes spontaneously or on command.
Recovery Time in PACU | Throughout the Post-Anesthesia Care Unit stay (up to 90 minutes)
  Time (minutes) spent in the PACU until Aldrete score ≥ 9.
Number of Patients Requiring Supplemental Propofol Boluses | During the gastroscopy procedure
  Count and percentage of patients requiring additional boluses of propofol after the initial induction dose.
Incidence of Respiratory Depression | From induction of anesthesia until emergence
  Percentage of patients experiencing respiratory depression (SpO2 < 90% for >30 seconds despite increased FiO2, apnea > 20 seconds, or signs of airway obstruction requiring intervention).
Incidence of Injection Pain | During intravenous drug administration at induction
  Percentage of patients experiencing bradycardia (heart rate decrease > 20% from baseline or below 5th percentile for age, especially if accompanied by hypotension or poor perfusion, requiring intervention).
Incidence of Postoperative Nausea and Vomiting (PONV) | Assessed in the Post-Anesthesia Care Unit and at 24 hours post-procedure
  Percentage of patients experiencing nausea or vomiting.
Incidence of Dizziness/Vertigo | Assessed in the Post-Anesthesia Care Unit and at 24 hours post-procedure
  Percentage of patients reporting dizziness or vertigo.
Satisfaction Scores | Assessed once at the time of discharge from the Post-Anesthesia Care Unit (PACU), which occurs approximately 30 to 90 minutes after the end of the procedure.
  Satisfaction levels of endoscopists, patients (if age ≥ 7 years and able to respond), and guardians, evaluated using a seven-point Likert scale (1 = very dissatisfied to 7 = very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Children's Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No